CLINICAL TRIAL: NCT04406012
Title: Analgesic Efficacy of Ultrasound Guided Paravertebral Block in Percutaneous Nephrolithotomy Patients: A Randomized Controlled Clinical Study
Brief Title: Analgesic Efficacy of Ultrasound Guided Paravertebral Block in Percutaneous Nephrolithotomy Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eskisehir Osmangazi University (Other)
Collaborators: Kırıkkale University (Other)
Responsible Party: Principal Investigator, Ferda YAMAN, Assist. Prof. Dr., Eskisehir Osmangazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Eskisehir University; Kırıkkale University (Other: No:04/03)
Record Dates: First submitted 2020-05-23; First posted 2020-05-28 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Pain, Postoperative; Anesthesia, Regional
Keywords: Pain management; Analgesia; paravertebral block; nephrolithotomy
MeSH Terms: conditions — Pain; Agnosia

STUDY DESIGN:
Intervention Model Description: Paravertebral block group and Control group
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- block group (Active Comparator): Paravertebral group at Thoracic 9-10 vertebrae level with an in-plane technique advanced ultrasound guided 10 ml bupivacaine hydrochloride (Marcaine 0.5%, Astra Zeneca) in 20 ml volume was enjected in the paravertebral area with real-time visualisation It was observed that the local anesthetic drug spread on the pleura and the pleura was pushed. All blocks were performed by the same experienced anaesthesiologist.
  Interventions: Procedure: paravertebral block
- Control group (No Intervention): Conventional analgesia methods were applied to the control group. Control group was relieved by dexketoprofen 50mg intravenously. If the patient was not relieved with dexketoprofen and VAS score >4, tramadol 1 mg kg-1 was administered intravenously.

INTERVENTIONS:
Procedure: paravertebral block — paravertebral block group
  Arms: block group

SUMMARY:
The aim of this study is to investigate the analgesic effects of thoracal paravertebral block in the patients undergoing percutaneous nephrolitotomy. Paravertebral block was applied to the study group. Conventional analgesia methods were applied to the control group.

DETAILED DESCRIPTION:
Randomization was divided into two groups by using closed envelope method. Postoperative pain scores at rest at 1, 2, 4, 6, 8, 10, 12, and 24 hours with VAS (0 = no pain, very severe pain = 10) using Visual Analogue Scale was made. VAS at rest and movement (coughing and taking a deep Breath) were evaluated. Patients with VAS> 4 received additional analgesics.

ELIGIBILITY:
ASA I, II, III patients aged 18-65 who consented to undergo unilateral percutaneous nephrolithotomy were eligible for the study. 53 patients were eligible and assesed.Informed consent was signed by all patients. Patients under 18 years of age, pregnant, with known hypersensitivity to local anesthetics, bleeding diathesis, depression and / or anxiety disorder, obesity (BMI> 35kg / m2), history of pneumothorax, phrenic nerve paralysis, severe aortic stenosis were excluded. Also who did not want to participate the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2016-02-16 (Actual); Primary Completion 2016-06-16 (Actual); Study Completion 2016-07-01 (Actual)

PRIMARY OUTCOMES:
Patient VAS scores | 24 hours
  0=no pain, 10=incredible pain

SECONDARY OUTCOMES:
Patient Satisfaction scores | at the end of the 24 hours
  0=not satisfied, 5=very good satisfied

IPD SHARING:
Plan to Share IPD: No
when the article published

REFERENCES:
- [Derived] Yaman F, Tuglu D. Analgesic efficacy of ultrasound guided paravertebral block in percutaneous nephrolithotomy patients: a randomized controlled clinical study. BMC Anesthesiol. 2020 Sep 29;20(1):250. doi: 10.1186/s12871-020-01169-6. PMID 32993528